CLINICAL TRIAL: NCT03576781
Title: Developing Brain Stimulation as a Treatment for Pain in Opiate Dependent Individuals: Parametric Assessment of 2 Evidence-based Strategies
Brief Title: Developing rTMS Treatment Strategies for Pain in Opiate Dependence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: South Carolina Clinical & Translational Research Institute (SCTR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 61328
Record Dates: First submitted 2018-06-12; First posted 2018-07-03 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Pain; Chronic Pain; Opioid Dependence; Opioid Use
Keywords: Brain Stimulation; Treatment
MeSH Terms: conditions — Pain; Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real iTBS to the DLPFC (Experimental): One session of real intermittent Theta Burst Stimulation (iTBS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC) (20 trains of stimulation over dlPFC (middle frontal gyrus) (F3); each train: 3 pulse bursts presented at 5Hz, 15 pulses/sec for 2 sec, 8 sec rest, 200 pulses/train; 110% RMT, MagPro; 600 pulses total)
  Interventions: Device: Real iTBS
- Sham iTBS to the DLPFC (Sham Comparator): One session of sham intermittent Theta Burst Stimulation (iTBS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC) (20 trains of stimulation over dlPFC (middle frontal gyrus) (F3); each train: 3 pulse bursts presented at 5Hz, 15 pulses/sec for 2 sec, 8 sec rest, 200 pulses/train; 110% RMT, MagPro; 600 pulses total)
  Interventions: Device: Sham iTBS
- Real cTBS to the MPFC (Experimental): One session of real continuous Theta Burst Stimulation (cTBS) will be delivered to the left medial prefrontal cortex (mPFC) (1 train of stimulation over the left frontal pole (FP1); each train: 3 pulse bursts presented at 5Hz, 15 pulses/sec for 40 sec, 600 pulses/train, 110% RMT, MagPro; 600 pulses total)
  Interventions: Device: Real cTBS
- Sham cTBS to the MPFC (Sham Comparator): One session of sham continuous Theta Burst Stimulation (cTBS) will be delivered to the left medial prefrontal cortex (mPFC) (1 train of stimulation over the left frontal pole (FP1); each train: 3 pulse bursts presented at 5Hz, 15 pulses/sec for 40 sec, 600 pulses/train, 110% RMT, MagPro; 600 pulses total)
  Interventions: Device: Sham cTBS

INTERVENTIONS:
Device: Real iTBS — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key)
  Arms: Real iTBS to the DLPFC
Device: Sham iTBS — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham iTBS to the DLPFC
Device: Real cTBS — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key).
  Arms: Real cTBS to the MPFC
Device: Sham cTBS — This will be delivered with the Magventure Magpro system; 600 pulses with the active sham coil (double blinded using the USB key). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham cTBS to the MPFC

SUMMARY:
The purpose of this study is to parametically evaluate two different types of repetitive Transcranial Magnetic Stimulation (rTMS) treatment strategies as a potential treatment for pain in individuals currently taking prescription opiates. Repetitive TMS is a non-invasive tool that uses magnetic pulses to temporarily stimulate specific brain areas. This study will test whether rTMS over different locations of the prefrontal cortex can produce a reduction in an individuals perception of pain and how the brain responds to pain. Participants will be randomized to receive either sham-rTMS, or one of two real rTMS treatments. Brain imaging, behavioral assessments, and pain assessments will be collected both immediately before and after rTMS.

DETAILED DESCRIPTION:
Chronic use of opiates is a rapidly escalating crisis in the United States, with over 4.3 million Americans dependent on opiate analgesic, an escalating rate of opiate overdose deaths, and a resurgence of intravenous heroin use leading to total societal cost exceeding $55 billion. The struggle to break the addiction cycle is likely due to factors that affect neural circuits that govern craving and cognitive control. There is growing interest in the utilization of prefrontal cortex repetitive transcranial magnetic stimulation (rTMS) as a novel, non-invasive, non-pharmacologic approach to decreasing craving among chronic opiate users. At this early stage of development, however, it is unclear if the best TMS strategy is to (Strategy 1, Aim 1) increase activity in the dorsolateral prefrontal cortex, or (Strategy 2, Aim 2) decrease activity in the ventromedial prefrontal cortex.

DESIGN: To parametrically evaluate these two promising treatment strategies, the investigators have developed a design where opiate dependent individuals and healthy controls will be randomized to receive either one placebo-like TMS treatment, or one of two real TMS treatments (DLPFC iTBS or MPFC cTBS). Participants with opiate dependence will be recruited from the local community, as well as the MUSC Center for Drug and Alcohol Programs (CDAP), the Ralph H. Johnson Substance Abuse Treatment Center and local pain clinics. Healthy controls will be recruited from the local community. Approved Study Team Members will visit the above mentioned clinics and community and talk with patients. Individuals who consent will receive interleaved TMS/BOLD imaging and our established MRI-based thermal pain paradigm immediately before and after rTMS. The investigators will also measure subjective pain and opiate craving ratings. The relative efficacy of Strategy 1 vs 2 will directly translate to development of a large clinical trial of rTMS as an innovative, new treatment option for pain in opiate dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand questionnaires and informed consent.
2. Able to read and understand questionnaires and informed consent.
3. Lives within 50 miles of the study site.
4. Is not at elevated risk of seizure (i.e., does not have a history of seizures, is not currently prescribed medications known to lower seizure threshold)
5. Does not have metal objects in the head/neck.
6. Does not have a history of traumatic brain injury, including a head injury that resulted in hospitalization, loss of consciousness for more than 10 minutes, or having ever been informed that they have an epidural, subdural, or subarachnoid hemorrhage.
7. Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

1. Any psychoactive illicit substance use (except marijuana and nicotine) within the last 30 days by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine THC levels.
2. Meets DSM IV criteria for current axis I disorders of major depression, panic disorder, obsessive-compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders, eating disorders, and any other psychotic disorder or organic mental disorder.
3. Has current suicidal ideation or homicidal ideation.
4. Has the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for ADHD.
5. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
6. Has current charges pending for a violent crime (not including DUI related offenses).
7. Does not have a stable living situation.
8. Suffers from chronic migraines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
iTBS to the left DLPFC vs. cTBS to the left MPFC | Day 1
  The effect of real vs. sham iTBS to the left DLPFC vs. real vs. sham cTBS to the left MPFC as a tool to modulate the brain response to pain will be assessed by comparing the brain activity in the executive circuit and limbic circuit before and after TMS.

SECONDARY OUTCOMES:
Changes in pain threshold | Day 1
  The Quantitative Sensory pain assessment produces 3 output variables: sensory threshold, pain threshold, tolerance threshold (expressed in degrees Celsius). The pain thresholds for individuals that receive both DLPFC and MPFC will be tested using a within subject repeated measures design (time x treatment) wherein time is the repeated variable and Real or Sham TMS is the grouping variable.
Changes in opiate pain and craving inventory | Day 1
  The Opiate Pain and Craving inventory produces 4 output variables of interest: level of discomfort, level of pain, urge to use opiates, amount willing to pay for an opiate. This will be tested using a within subject repeated measures design (time x treatment) wherein time is the repeated variable and Real or Sham TMS is the grouping variable.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Ralph H Johnson Veterans Medical Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. All data is deidentified.